CLINICAL TRIAL: NCT00226980
Title: A Phase II Trial of Thalidomide and Capecitabine in Metastatic Renal Cell Carcinoma
Brief Title: A Trial of Thalidomide and Capecitabine in Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sandy Srinivas, Principal Investigator, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENAL0001; NCT00226980; RENAL0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Thalidomide; Capecitabine

INTERVENTIONS:
Drug: Thalidomide
Drug: Capecitabine

SUMMARY:
The purpose of this study is to determine the efficacy of the combination of thalidomide and capecitabine in metastatic renal cell carcinoma and also to determine the safety of the combination.

ELIGIBILITY:
Inclusion Criteria:- Able to comprehend and sign an IRB approved Informed consent

* Willingness and ability to comply with the FDA-mandated S.T.E.P.S.® program.
* Male or female 18 years or older
* Willing to use contraception
* Pathologic diagnosis of renal cell carcinoma
* Bi-dimensionally measurable disease
* Evidence of disease progression prior to start of treatment
* Failed prior immunotherapy or unwilling/unable to receive prior immunotherapy
* Adequate hematologic data: ANC.1.5; platelets>100x10^9
* Adequate renal function: Creatinine clearance .50cc
* Adequate liver function: Alkaline phos <3XULN AST/ALT <3XULN T.Bili <1.5XULN
* ECOG performance status 0-1 Exclusion Criteria:- Known brain metastases.
* Peripheral neuropathy.
* Pregnant and/ or lactating female.
* Unable to take a baby aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-10; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the combination of thalidomide and capecitabine in metastatic renal cell carcinoma.

SECONDARY OUTCOMES:
Safety of the combination

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States